CLINICAL TRIAL: NCT04875663
Title: Enhancing Group Lifestyle Intervention for Depression With Self-Tracking Tools: A Randomized Controlled Trial
Brief Title: Enhancing Group Lifestyle Intervention for Depression With Self-Tracking Tools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY015
Record Dates: First submitted 2021-05-05; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Depression
Keywords: Lifestyle medicine; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle medicine intervention with self-tracking tools (Experimental): Lifestyle intervention including diet, sleep, exercise, relaxation, and mindfulness. Self-tracking tools including a smartphone application and an Actigraphy will be given.
  Interventions: Behavioral: Lifestyle Medicine
- Pure lifestyle medicine intervention (Experimental): Lifestyle intervention including diet, sleep, exercise, relaxation, and mindfulness.
  Interventions: Behavioral: Lifestyle Medicine
- Care-As-Usual (No Intervention): continue receiving the routine care as usual and be given a smartphone-based LM intervention after the completion of follow-up assessments

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle intervention including diet, sleep, exercise, relaxation and mindfulness
  Arms: Lifestyle medicine intervention with self-tracking tools; Pure lifestyle medicine intervention

SUMMARY:
This study will be a randomized controlled trial on the effects of group-based LM as an intervention for depression. Prior to all study procedures, an online informed consent (with phone support) will be obtained from potential participants. Around 90 eligible participants will be randomly assigned to either the LM intervention with self-tracking tools (LM/S), pure LM intervention (LM), or care-as-usual (CAU) control group in a ratio of 1:1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. In order to obtain unbiased data with respect to the participants' attitudes and behaviors, incomplete disclosure will be used to withhold the self-tracking component in this trial. Participants in the two LM groups will receive six weekly group lifestyle modification sessions (~2 hours each) at the Chinese University of Hong Kong (an online approach will be adopted if face-to-face sessions are not possible due to COVID-19). The group treatment will primarily be delivered by clinical psychology trainees under the supervision of a clinical psychologist and other healthcare professionals such as a dietitian and a fitness trainer. The CAU group will continue receiving the routine care as usual and be given a smartphone-based LM intervention after the completion of follow-up assessments. Both the treatment groups and control group will complete a set of online questionnaires before the treatment commences, immediately after treatment, and 12 weeks after the treatment sessions are completed. In addition, participants in the LM/S group will complete a set of self-developed survey questions related to lifestyle and mood on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged ≥ 18 years
2. Cantonese language fluency and readability
3. A Patient Health Questionnaire 9 items (PHQ-9) score of at least 10, indicating a moderate level of depression
4. Possession of an internet-enabled mobile device (iOS or Android operating system)
5. Willingness to provide informed consent and comply with the trial protocol

Exclusion Criteria:

1. Current serious suicidal risk (non-fleeting intent or plan) as assessed by a PHQ-9 Item 9 score > 2 (referral information to professional mental health services will be provided)
2. Any medical or neurocognitive disorder(s) that makes participation unsuitable based on the team's clinical experience or interferes with adherence to the lifestyle modification (e.g., where exercise or a change in diet are not recommended by physicians)
3. Current involvement in lifestyle changes supervised by professionals
4. Unstable medication or current participation in any psychotherapy for depression
5. Pregnancy
6. Hospitalization
7. Current participation in any other trial(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  The GAD-7, a 7-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of anxiety over the past two weeks on a 4-point scale, "0" (not at all) to "4" (nearly every day).
Change in Insomnia Severity Index (ISI) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the World Health Organization Quality of Life Instruments (WHOQOL-BREF) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  WHOQOL-BREF consists of 24 items assessing perception of quality of life (QoL) in four domains, including physical health, psychological, social relationships, and environment, and two items on overall QoL and general health. The domain scores were transformed into a linear scale between 0 and 100 following the scoring guidelines. A higher score indicated a better QoL.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from a short form of the International Physical Activity Questionnaire - Chinese version a short form of the IPAQ-C.

OTHER OUTCOMES:
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediately after treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong